CLINICAL TRIAL: NCT02841527
Title: Gastric Bypass, Adjustable Gastric Banding or Sleeve Gastrectomy Surgery to Treat Severe and Complex Obesity: a Multi-centre Randomised Controlled Trial
Brief Title: Gastric Bypass, Gastric Band or Sleeve Gastrectomy to Treat Obesity
Acronym: ByBandSleeve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bristol (Other)
Collaborators: University of Oxford (Other); University of Birmingham (Other)
Responsible Party: Principal Investigator, Jane Blazeby, Chief Investigator, University of Bristol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORCA39300
Record Dates: First submitted 2016-04-08; First posted 2016-07-22 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Surgery; Quality of Life; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gastric Band (Active Comparator): The procedure will involve an operation in which a gastric Band and port will be fitted using a laparoscopic technique.
  Interventions: Procedure: Gastric Band
- Gastric Bypass (Active Comparator): The procedure will involve a laparoscopic operation in which a small pouch is made in the top of the stomach and a loop of bowel connected to this pouch to bypass the rest of the stomach.
  Interventions: Procedure: Gastric Bypass
- Sleeve Gastrectomy (Active Comparator): The procedure involves an operation which reduces the size of the stomach by about 75%, creating a narrow tube. It is done by stapling down the stomach and removing the remainder of the stomach using a laparoscopic technique.
  Interventions: Procedure: Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Gastric Band — Surgical intervention in which a band is inserted around the top of the stomach to reduce its size.
  Arms: Gastric Band
Procedure: Gastric Bypass — Surgical intervention where a small pouch is made in the top of the stomach and a loop of bowel connected to this pouch to bypass the rest of the stomach.
  Arms: Gastric Bypass
Procedure: Sleeve Gastrectomy — Surgical intervention which reduces the size of the stomach by about 75%, creating a narrow tube. It is done by stapling down the stomach and removing the remainder of the stomach.
  Arms: Sleeve Gastrectomy

SUMMARY:
Obesity is an increasing health problem in the United Kingdom (UK) and is predicted to worsen.

In the UK and worldwide the three most commonly performed operations are laparoscopic adjustable gastric banding ('BAND surgery'), laparoscopic gastric bypass ('BYPASS') and laparoscopic sleeve gastrectomy ('SLEEVE'). All lead to weight loss, but they are associated with different problems. This study (BYBANDSLEEVE) is a randomised trial with a target recruitment of 1341 patients in twelve hospitals and its aim is to compare the effectiveness, cost effectiveness and acceptability of BAND, BYPASS and SLEEVE surgery.

DETAILED DESCRIPTION:
Obesity is an increasing health problem in the UK and one which is predicted to worsen. It is associated with many health problems that can shorten a person's life span and impair quality of life. Current national guidelines recommend that surgery is considered for the very overweight (morbidly obese) or for those remaining obese after trying other options.

In the UK and worldwide the three most commonly performed operations are laparoscopic adjustable gastric banding ('BAND surgery'), laparoscopic gastric bypass ('BYPASS') and laparoscopic sleeve gastrectomy ('SLEEVE'). All lead to weight loss, but they are associated with different problems. In the short term there are varying complications and inconvenience relating to the operation. In the longer term there are different outcomes relating to weight regain, symptoms and side effects of surgery. This study (BYBANDSLEEVE) is a randomised trial with a recruitment target of 1341 patients in twelve hospitals and its aim is to compare the effectiveness, cost effectiveness and acceptability of BAND, BYPASS and SLEEVE surgery. The process of randomisation will mean that participants have a chance of receiving one of the three procedures, so a fair comparison between them can be made.

The first phase (in two hospitals) will test the feasibility of recruitment and optimise information for patients to maximise trial recruitment. It will establish a core set of clinical outcomes to use to evaluate the surgery for morbid obesity. The second stage (in 12 hospitals) will recruit the full sample and follow up all participants for at least three years. The investigators will compare the effects of BAND, BYPASS AND SLEEVE surgery three years after randomisation on weight loss, a wide range of symptoms and aspects of quality of life. The investigators will also examine patients' detailed experiences during follow up, nutritional outcomes, short and long term surgical complications and National Health Service (NHS) value for money.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients
2. Over 18 years of age
3. Referred for bariatric surgery according to the National Institute for Health and Care Excellence (NICE) guidelines - BMI of 40kg/m2 or more, OR BMI of 35 kg/m2 to 40 kg/m2 and other significant disease (e.g. type 2 diabetes or high blood pressure) OR BMI of 30 kg/m2 or more and recent onset diabetes OR Asian family origin with lower BMI and recent onset diabetes, that could improve with weight loss
4. Has been or is willing to receive intensive management in a specialist tier 3 obesity service
5. Fit for anaesthesia and surgery
6. Committed to follow-up and able to complete quality of life questionnaires
7. Able to provide written informed consent.

Exclusion Criteria:

1. Previous gastric surgery or surgery for severe and complex obesity
2. Previous abdominal surgery or gastro-intestinal (GI) condition that precludes one or more of Band, Bypass or Sleeve
3. Large abdominal ventral hernia
4. Pregnancy (women who have given birth and women planning pregnancy will NOT be excluded)
5. Crohn's disease
6. Liver cirrhosis and portal hypertension
7. Systemic lupus erythematosis
8. Known silicone allergy
9. Hiatus hernia >5cm
10. Other clinical/psychological reason, to be specified
11. Active participation in another interventional research study which might interfere with By-Band-Sleeve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1351 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The proportion achieving loss of greater than 50% of excess weight at three years. | Three years
  The proportion achieving loss of greater than 50% of excess weight at three years (calculated as 100×[BMI at 3 years - BMI at randomisation1] / [BMI at randomisation - 25])
Health-related Quality of Life (HRQoL) | Three years
  HRQoL at three 3 years, will be assessed using the EQ-5D-5L

SECONDARY OUTCOMES:
Change in BMI over time adjusted for BMI at randomisation | Three years
  Change in BMI over time adjusted for BMI at randomisation
Percentage weight loss at 3 years | Three years
  Percentage weight loss at 3 years
Waist circumference at 3 years | Three years
  Waist circumference at 3 years
Time taken from randomisation to reach first loss of at least 50% of excess BMI | Three years
  Time taken from randomisation to reach first loss of at least 50% of excess BMI
Time taken from first losing 50% excess BMI to first relapse | Three years
  Time taken from first losing 50% excess BMI to first relapse (defined as weight re-gain such that the target of at least 50% of excess weight loss is no longer met)
Generic and symptom specific Health-related Quality of Life (HRQOL) | Three years
  Impact of Weight on Quality of Life (IWQOL-Lite)
Generic and symptom specific Health-related Quality of Life (HRQOL) | Three years
  The Gastrointestinal Quality of Life Index
Generic and symptom specific Health-related Quality of Life (HRQOL) | Three years
  Eating Habits Questionnaire
Generic and symptom specific Health-related Quality of Life (HRQOL) | Three years
  SF-12v2 Health Survey
Generic and symptom specific Health-related Quality of Life (HRQOL) | Three years
  Hospital Anxiety and Depression Scale (HADS).
Resource use to three years | Three years
  Use of health service resources over the three-year study period.
Standard healthcare blood tests | Three years
  Standard NHS nutritional blood tests will be performed at each assessment.
Dietary recall | Three years
  Measures of 24 hour recall eating using a standardised and validated interview process
Binge eating behaviour | Three years
  Binge eating behaviour using a validated questionnaire
Adverse health events | Three years
  Adverse health events including the need for re-operation and cross over between interventions
Resolution of co-morbidities | Three years
  Resolution of co-morbidities at 3 years, including sleep apnoea, non alcoholic fatty liver disease, type-2 diabetes, hypertension and hyperlipidaemia.
Time to resolution of co-morbidities | Three years
  Time to resolution of sleep apnoea, type-2 diabetes, hypertension and hyperlipidaemia

CONTACTS AND LOCATIONS:
Overall Officials: Jane Blazeby, BSc,MBChB,MD, Study Director — University of Bristol
Locations (12):
- United Kingdom (12):
  - Heart of England NHS Foundation Trust, Birmingham
  - Royal Bournemouth and Christchurch Hospitals, Bournemouth
  - North Bristol NHS Trust, Bristol
  - Royal Derby Hospital, Derby
  - St James University Hospital, Leeds, Leeds
  - Homerton University Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Queen Alexandra Hospital, Portsmouth
  - University Hospital Southampton, Southampton
  - Sunderland Royal Hospital, Sunderland
  - Musgrove Park Hospital, Taunton
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No
All data will be anonymised and analysed in groups. Individual patient data (IPD) will be made available to the research team following analysis.

REFERENCES:
- [Background] Blazeby JM, Byrne J, Welbourn R. What is the most effective operation for adults with severe and complex obesity? BMJ. 2014 Mar 14;348:g1763. doi: 10.1136/bmj.g1763. No abstract available. PMID 24633209
- [Background] Donovan JL, Paramasivan S, de Salis I, Toerien M. Clear obstacles and hidden challenges: understanding recruiter perspectives in six pragmatic randomised controlled trials. Trials. 2014 Jan 6;15:5. doi: 10.1186/1745-6215-15-5. PMID 24393291
- [Background] Rogers CA, Welbourn R, Byrne J, Donovan JL, Reeves BC, Wordsworth S, Andrews R, Thompson JL, Roderick P, Mahon D, Noble H, Kelly J, Mazza G, Pike K, Paramasivan S, Blencowe N, Perkins M, Porter T, Blazeby JM. The By-Band study: gastric bypass or adjustable gastric band surgery to treat morbid obesity: study protocol for a multi-centre randomised controlled trial with an internal pilot phase. Trials. 2014 Feb 11;15:53. doi: 10.1186/1745-6215-15-53. PMID 24517309
- [Background] Hopkins JC, Howes N, Chalmers K, Savovic J, Whale K, Coulman KD, Welbourn R, Whistance RN, Andrews RC, Byrne JP, Mahon D, Blazeby JM; By-Band Trial Management Group. Outcome reporting in bariatric surgery: an in-depth analysis to inform the development of a core outcome set, the BARIACT Study. Obes Rev. 2015 Jan;16(1):88-106. doi: 10.1111/obr.12240. Epub 2014 Nov 30. PMID 25442513
- [Background] Coulman KD, Hopkins J, Brookes ST, Chalmers K, Main B, Owen-Smith A, Andrews RC, Byrne J, Donovan JL, Mazza G, Reeves BC, Rogers CA, Thompson JL, Welbourn R, Wordsworth S, Blazeby JM; BARIACT working group. A Core Outcome Set for the Benefits and Adverse Events of Bariatric and Metabolic Surgery: The BARIACT Project. PLoS Med. 2016 Nov 29;13(11):e1002187. doi: 10.1371/journal.pmed.1002187. eCollection 2016 Nov. PMID 27898680
- [Background] Coulman KD, Howes N, Hopkins J, Whale K, Chalmers K, Brookes S, Nicholson A, Savovic J, Ferguson Y, Owen-Smith A, Blazeby J; By-Band-Sleeve Trial Management Group; Blazeby J, Welbourn R, Byrne J, Donovan J, Reeves BC, Wordsworth S, Andrews R, Thompson JL, Mazza G, Rogers CA. A Comparison of Health Professionals' and Patients' Views of the Importance of Outcomes of Bariatric Surgery. Obes Surg. 2016 Nov;26(11):2738-2746. doi: 10.1007/s11695-016-2186-0. PMID 27138600
- [Background] Hopkins JC, Blazeby JM, Rogers CA, Welbourn R. The use of adjustable gastric bands for management of severe and complex obesity. Br Med Bull. 2016 Jun;118(1):64-72. doi: 10.1093/bmb/ldw012. Epub 2016 Mar 31. PMID 27034443
- [Background] Rooshenas L, Elliott D, Wade J, Jepson M, Paramasivan S, Strong S, Wilson C, Beard D, Blazeby JM, Birtle A, Halliday A, Rogers CA, Stein R, Donovan JL; ACST-2 study group; By-Band-Sleeve study group; Chemorad study group; CSAW study group; Optima prelim study group; POUT study group. Conveying Equipoise during Recruitment for Clinical Trials: Qualitative Synthesis of Clinicians' Practices across Six Randomised Controlled Trials. PLoS Med. 2016 Oct 18;13(10):e1002147. doi: 10.1371/journal.pmed.1002147. eCollection 2016 Oct. PMID 27755555
- [Background] Welbourn R, le Roux CW, Owen-Smith A, Wordsworth S, Blazeby JM. Why the NHS should do more bariatric surgery; how much should we do? BMJ. 2016 May 11;353:i1472. doi: 10.1136/bmj.i1472. No abstract available. PMID 27169605
- [Background] Doble B, Wordsworth S, Rogers CA, Welbourn R, Byrne J, Blazeby JM; By-Band-Sleeve Trial Management Group. What Are the Real Procedural Costs of Bariatric Surgery? A Systematic Literature Review of Published Cost Analyses. Obes Surg. 2017 Aug;27(8):2179-2192. doi: 10.1007/s11695-017-2749-8. PMID 28550438
- [Background] Fermont JM, Blazeby JM, Rogers CA, Wordsworth S; By-Band-Sleeve Study Management Group. The EQ-5D-5L is a valid approach to measure health related quality of life in patients undergoing bariatric surgery. PLoS One. 2017 Dec 18;12(12):e0189190. doi: 10.1371/journal.pone.0189190. eCollection 2017. PMID 29252996
- [Background] Paramasivan S, Rogers CA, Welbourn R, Byrne JP, Salter N, Mahon D, Noble H, Kelly J, Mazza G, Whybrow P, Andrews RC, Wilson C, Blazeby JM, Donovan JL. Enabling recruitment success in bariatric surgical trials: pilot phase of the By-Band-Sleeve study. Int J Obes (Lond). 2017 Nov;41(11):1654-1661. doi: 10.1038/ijo.2017.153. Epub 2017 Jul 3. PMID 28669987
- [Background] Rogers CA, Reeves BC, Byrne J, Donovan JL, Mazza G, Paramasivan S, Andrews RC, Wordsworth S, Thompson J, Blazeby JM, Welbourn R; By-Band-Sleeve study investigators. Adaptation of the By-Band randomized clinical trial to By-Band-Sleeve to include a new intervention and maintain relevance of the study to practice. Br J Surg. 2017 Aug;104(9):1207-1214. doi: 10.1002/bjs.10562. PMID 28703939
- [Background] Doble B, Welbourn R, Carter N, Byrne J, Rogers CA, Blazeby JM, Wordsworth S; By-Band-Sleeve Trial Management Group. Multi-Centre Micro-Costing of Roux-En-Y Gastric Bypass, Sleeve Gastrectomy and Adjustable Gastric Banding Procedures for the Treatment of Severe, Complex Obesity. Obes Surg. 2019 Feb;29(2):474-484. doi: 10.1007/s11695-018-3553-9. PMID 30368646
- [Background] Rooshenas L, Scott LJ, Blazeby JM, Rogers CA, Tilling KM, Husbands S, Conefrey C, Mills N, Stein RC, Metcalfe C, Carr AJ, Beard DJ, Davis T, Paramasivan S, Jepson M, Avery K, Elliott D, Wilson C, Donovan JL; By-Band-Sleeve study group; CSAW study group; HAND-1 study group; Optima prelim study group; Romio feasibility study group. The QuinteT Recruitment Intervention supported five randomized trials to recruit to target: a mixed-methods evaluation. J Clin Epidemiol. 2019 Feb;106:108-120. doi: 10.1016/j.jclinepi.2018.10.004. Epub 2018 Oct 16. PMID 30339938
- [Derived] Roux-en-Y gastric bypass, adjustable gastric banding or sleeve gastrectomy for severe obesity: The By-Band-Sleeve randomised controlled trial. Health Technol Assess. 2026 Jan;30(6):1-224. doi: 10.3310/CXSE2951. PMID 41631732
- [Derived] By-Band-Sleeve Collaborative Group. Roux-en-Y gastric bypass, adjustable gastric banding, or sleeve gastrectomy for severe obesity (By-Band-Sleeve): a multicentre, open label, three-group, randomised controlled trial. Lancet Diabetes Endocrinol. 2025 May;13(5):410-426. doi: 10.1016/S2213-8587(25)00025-7. Epub 2025 Mar 31. PMID 40179925
- [Derived] By-Band-Sleeve Collaborating Group. Prevalence and short-term change in symptoms of anxiety and depression following bariatric surgery: a prospective cohort study. BMJ Open. 2024 Jan 3;14(1):e071231. doi: 10.1136/bmjopen-2022-071231. PMID 38171620
- [Derived] By-Band-Sleeve Collaborative Group. Roux-en-Y gastric bypass, gastric banding, or sleeve gastrectomy for severe obesity: Baseline data from the By-Band-Sleeve randomized controlled trial. Obesity (Silver Spring). 2023 May;31(5):1290-1299. doi: 10.1002/oby.23746. PMID 37140395
- See also: By-Band-Sleeve study website — http://www.by-band-sleeve.bristol.ac.uk/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT02841527/Prot_SAP_001.pdf